CLINICAL TRIAL: NCT05835024
Title: A Multi-Site Observational Clinical Investigation to Collect Non-invasive Sensor Data During a Right Heart Catheterization and Train Machine Learning Models to Estimate Intracardiac Hemodynamic Parameters Evaluation of a Novel maChine leArning Model's Performance for Non-invasive inTracardiac pressURE Monitoring in Heart Failure - The CAPTURE-HF Trial
Brief Title: Acorai Machine Learning Generalization (MLG) Study
Acronym: CAPTURE-HF
Status: Completed | Type: Observational
Sponsor: Acorai AB (Industry)
Responsible Party: Sponsor
Other Study IDs: ASDC-1
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants phase 1: Phase 1: patients enrolled for a right heart catheterization procedure as part of their standard of care.
  Interventions: Device: Acorai Sensor Data Collection (ASDC) system 1.0 - Phase 1
- Participants phase 2: Phase 2: patients enrolled for a right heart catheterization procedure as part of their standard of care.
  Interventions: Device: Acorai Sensor Data Collection (ASDC) system 1.0 - Phase 2

INTERVENTIONS:
Device: Acorai Sensor Data Collection (ASDC) system 1.0 - Phase 1 — A supervised session that includes 10 minutes of patient information entry, 5 minutes of sensor recording time and 10 minutes of margin for setting up the system and patient, thus a total evaluation duration of approximately 25 minutes prior to the Right Heart Catheterization.
  No follow-up period for the subjects will be required for this clinical investigation. Patients will be followed as per standard of care, at the hospital.
  A single follow-up observational data collection will be conducted at 90 days, to collect the number of unplanned hospitalizations since the procedure visit. This does not involve active patient participation.
  Groups: Participants phase 1
Device: Acorai Sensor Data Collection (ASDC) system 1.0 - Phase 2 — A supervised session that includes 10 minutes of patient information entry, 5 minutes of sensor recording time and 10 minutes of margin for setting up the system and patient, thus a total evaluation duration of approximately 25 minutes prior to the Right Heart Catheterization.
  No follow-up period for the subjects will be required for this clinical investigation. Patients will be followed as per standard of care, at the hospital.
  Groups: Participants phase 2

SUMMARY:
Acorai is developing a non-invasive monitoring system for the estimation of intracardiac hemodynamic parameters in patients with suspected or confirmed heart failure, and/or pulmonary hypertension, who require hemodynamic assessment. The device will be intended as a companion test or clinical decision support tool to be used and interpreted by qualified healthcare professionals to aid standard-of-care clinical assessment in identifying hemodynamic congestion and supporting personalized treatment of heart failure and pulmonary congestion.

This study is part of the development of a non-invasive monitoring system for the estimation of intracardiac hemodynamic parameters. It will be conducted to collect the data needed to train the machine learning models retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Subject is, at least, 18 years of age at the time of screening visit.
* Subject is willing and physically able to comply with the specified evaluations as per the clinical investigation plan, as assessed by the investigator.
* Subject is referred for invasive hemodynamic assessment with right heart cardiac catheterization.
* Patient has provided written informed consent using the Ethics Committee/ Institutional Review Board approved consent form.

Exclusion Criteria:

* Discretionary exclusion when, in the opinion of the investigator, the inclusion of a potential subject is not in their best interest or not in the interest of compliant performance of the clinical investigation.
* Subjects who are pregnant are excluded in the US

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients enrolled for a right heart catheterization procedure as part of their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 1602 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the ML's performance to estimate pressure | Day 0 to Day 90
  Performance of the ML model trained on data collected from the ASDC System to estimate left-sided filling pressure compared to right heart catheterization.

SECONDARY OUTCOMES:
Evaluation of the ML's performance to estimate other hemodynamic parameters | Day 0 to Day 90
  The performance of the ML model trained on data collected from the ASDC System to estimate other hemodynamic parameters (such as right atrial pressure) compared to right heart catheterization.
Diagnostic accuracy of ML model | Day 0 to Day 90
  The diagnostic accuracy of the ML model trained on data collected from the ASDC System to detect clinically significant abnormal right heart catheterization measurements.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (10):
  - Conway Regional Cardiovascular Clinic, Conway, Arkansas
  - Baptist Health Medical Centre, Little Rock, Arkansas
  - Mayo Clinic, Jacksonville, Florida
  - Cleveland Clinic Martin Health, Stuart, Florida
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - WakeMed, Raleigh, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Austin Heart Central and San Marcos, Austin, Texas
  - Austin Heart Round Rock, Austin, Texas
- Onze-Lieve-Vrouwziekenhuis (OLV) Hospital Aalst, Aalst, Belgium
- Canada (3):
  - University of Ottawa Heart Institute, Ottawa
  - Mount Sinai Hospital Toronto, Toronto
  - Toronto General Hospital, Toronto
- Rigshospitalet, University Hospital of Copenhagen, Copenhagen, Denmark
- Sahlgrenska university hospital, Gothenburg, Sweden
- United Kingdom (2):
  - Royal Brompton and Harefield Hospitals, London
  - Southampton University Hospital, Southampton